CLINICAL TRIAL: NCT02175069
Title: Magnetic Resonance Imaging of Local Anesthetic Distribution: A Comparison of 5 and 15 Milliliters of Ropivacaine 0,75% for Ultrasound Guided Interscalene Plexus Blockade
Brief Title: Magnetic Resonance Imaging of Interscalene Plexus Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Prof. Peter Gerner, M.D., Prim. Univ.-Prof. Dr. med. univ. Peter Gerner, Paracelsus Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MR-ISB-1
Record Dates: First submitted 2014-04-17; First posted 2014-06-26 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Disorder of Shoulder
Keywords: Shoulder surgery
MeSH Terms: interventions — Ropivacaine; Gadolinium DTPA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interscalene Nerve Block - 5ml (Experimental): ultrasound guided interscalene plexus block (UISB)
  Ropivacaine 0.75%, 20ml Gadopentetate-Dimeglumine 0.05 mmol Shoulder Surgery
  Interventions: Procedure: Interscalene Nerve Block; Drug: Gadopentetate-Dimeglumine 0.0125 mmol; Drug: Ropivacaine 0.75%, 5ml; Procedure: Shoulder Surgery
- Interscalene Nerve Block - 20ml (Active Comparator): ultrasound guided interscalene plexus block (UISB)
  Ropivacaine 0.75%, 5ml Gadopentetate-Dimeglumine 0.0125 mmol Shoulder Surgery
  Interventions: Procedure: Interscalene Nerve Block; Drug: Ropivacaine 0.75%, 20ml; Drug: Gadopentetate-Dimeglumine 0.05 mmol; Procedure: Shoulder Surgery

INTERVENTIONS:
Procedure: Interscalene Nerve Block — ultrasound guided interscalene plexus block (UISB) immediately before magnetic resonance imaging of the neck.
Drug: Ropivacaine 0.75%, 20ml — 20 ml of ropivacaine 0.75%
  Other Names: Naropin
  Arms: Interscalene Nerve Block - 20ml
Drug: Gadopentetate-Dimeglumine 0.0125 mmol — 0.0125 mmol of gadopentetate-dimeglumine
  Other Names: Magnevist
  Arms: Interscalene Nerve Block - 5ml
Drug: Gadopentetate-Dimeglumine 0.05 mmol — 0.05 mmol of gadopentetate-dimeglumine
  Other Names: Magnevist
  Arms: Interscalene Nerve Block - 20ml
Drug: Ropivacaine 0.75%, 5ml — 5 ml of ropivacaine 0.75%
  Other Names: Naropin
  Arms: Interscalene Nerve Block - 5ml
Procedure: Shoulder Surgery — As per individual requirement (patient-dependent)

SUMMARY:
Interscalene plexus block is a widely used technique to provide anesthesia and analgesia for surgery at the upper extremity (shoulder and upper arm); it is standard-of-care in many institutions worldwide. Local anesthetic is being injected around the nerves supplying the arm (Plexus brachialis) at a specific location in the arm (between the scalenus muscles, thus called "interscalene plexus block"). The optimal volume of injection with regard to efficacy, safety and avoidance of untoward effects has been subject to intense debate for a long time. In spite of evidence that small volumes (between 5 and 7 mls) are effective for adequate postoperative analgesia, larger volumes up to 40 mls are still frequently used in many practices. However, with the use of such large doses, adverse events are known to occur with increased frequency, including paralysis of the diaphragm or spread of local anesthetic to the spinal cord.

This study is intended to help evaluate the effects of small or larger injection of local anesthetic around the brachial plexus, and to correlate the distribution with clinical efficacy, block duration, and possible side effects. It is a randomized, controlled, observer-blinded trial; patients undergoing shoulder or upper arm surgery will be randomly allocated to receive either 5mls or 20mls of local anesthetic for their interscalene plexus block. Magnetic resonance imaging will be performed immediately afterwards, followed by a series of neurological exams during the hospital stay. Test of lung function (spirometry) and ultrasound of the diaphragm will be used to evaluate effects of the block on respiratory mechanics.

DETAILED DESCRIPTION:
Background: Interscalene plexus blockade (ISB) is frequently used during surgery of the upper limb. The use of ultrasound has significantly reduced time of onset and total volume of local anesthetics in comparison to nerve localization by stimulators. (1-4) The introduction of this technique has been correlated with decreased volumes of effective local anesthetics from 40 milliliters and more down to 10 milliliters and less.(3-4) As the injection site of ISB is located in close proximity to the anatomical structures of the spinal cord, spread of local anesthetics could potentially cause adverse events, including contralateral blockade and total spinal anesthesia. Case reports on these complications have been published previously. (5-11)In a recently published study we showed that the phenomenon of epidural spread can be reproduced in cadavers and seems to be positively correlated to injection-volumes exceeding 10 milliliters.(12) Moreover, we observed a trend towards cranial spread of the contrast agent in all investigated specimens along the course of the nerval roots towards the spinal cord. In another cadaveric study by Orebauch et al., cranial epidural spread was also detectable following injection of dye into the nerval roots of the brachial plexus.(13) Magnetic resonance imaging has not yet been used for visualization of the spread of local anaesthetics in ISB.

Given that ultrasound provides excellent visualization of target-structures in regional anesthesia and therefore enables physicians to place injection needles with enormous accuracy, the question arises whether there is a critical volume for local anesthetics increasing complications such as epidural spread and in consequence contralateral blockade.

The aim of this study is to confirm the findings of our cadaveric study in vivo and to show that the frequency of epidural spread correlates with injection of increased volumes of local anesthetics.

Primary endpoint: Spread of local anesthetics to the epidural space

Secondary endpoints:

* Contralateral epidural spread.
* Spread of local anesthetics to the phrenic nerve.
* Bed side spirometry and ultrasound investigation of the diaphragm in the PACU.
* Oxygen saturation in the PACU
* Self-reported block duration.
* Self reported pain scores for the first 24 postoperative hours
* Time to first analgesic consumption on demand.
* Total analgesic consumption (ropivacaine PCA).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Surgery of the shoulder (shoulder arthroscopy, open shoulder joint surgery, rotator cuff surgery, tendon transfer, shoulder arthroplasty, humerus fracture surgery)
* Patients willing to undergo magnetic resonance imaging prior to surgery
* Informed consent to participate in the study
* American Society of Anesthesiologists physical score I, II or III

Exclusion Criteria:

* Refusal to participate in the study
* Inability to understand the study protocol due to language barrier
* Serious cardiac or pulmonary disease such as decompensated heart failure, recent myocardial infarction (less than one month in the past), heart block greater than 2nd degree, obstructive sleep apnea and chronic obstructive lung disease greater than 2nd degree
* renal impairment with an calculated glomerular filtration rate below 60ml/min
* Hypersensitivity to ropivacaine or gadolinium or other contraindications against peripheral nerve blocks
* Chronic opioid usage greater than 15 mg oral morphine equivalents daily, the daily use of adjunctive pain medications (gabapentins, tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitors)
* Schizophrenia or bipolar disorders, uncontrolled anxiety, claustrophobia
* Peripheral neuropathy
* Hepatic or renal impairment
* Ongoing illicit drug or alcohol abuse
* Metal implants or other contraindications for magnetic resonance imaging
* Coagulopathy
* Participation in additional clinical trials within 4 weeks before screening
* Hearing impairment
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Spread of local anesthetics to the epidural space | 10 minutes
  Spread of local anesthetics to the epidural space, as seen in the magnetic resonance imaging

SECONDARY OUTCOMES:
Contralateral epidural spread | 10 min
  as seen on MRI
Spread of local anesthetics to the phrenic nerve | 10 minutes
  as seen on MRI
Bed side spirometry and ultrasound investigation of the diaphragm in the PACU | 24 hours
Oxygen saturation in the PACU | 2-6 hours
Self-reported block duration | 24 hours
Self reported pain scores for the first 24 postoperative hours | 24 hrs
Time to first analgesic consumption on demand | 24 hours
Total analgesic consumption (ropivacaine PCA). | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gerner, MD, Study Chair — Department of Anesthesiology, Perioperative Medicine and Intensive Care, Paracelsus Medical University, Salzburg, Austria; Gerhard Fritsch, MD, Principal Investigator — Department of Anesthesiology, Perioperative Medicine and Intensive Care, Paracelsus Medical University, Salzburg, Austria
Locations (1):
- Paracelsus Medical University, Department of Anesthesiology, Salzburg, Salzburg, Austria

REFERENCES:
- [Background] Fredrickson MJ, Ball CM, Dalgleish AJ. A prospective randomized comparison of ultrasound guidance versus neurostimulation for interscalene catheter placement. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):590-4. doi: 10.1097/aap.0b013e3181ada622. PMID 19916253
- [Background] Fredrickson MJ, Ball CM, Dalgleish AJ, Stewart AW, Short TG. A prospective randomized comparison of ultrasound and neurostimulation as needle end points for interscalene catheter placement. Anesth Analg. 2009 May;108(5):1695-700. doi: 10.1213/ane.0b013e31819c29b8. PMID 19372356
- [Background] Gautier P, Vandepitte C, Ramquet C, DeCoopman M, Xu D, Hadzic A. The minimum effective anesthetic volume of 0.75% ropivacaine in ultrasound-guided interscalene brachial plexus block. Anesth Analg. 2011 Oct;113(4):951-5. doi: 10.1213/ANE.0b013e31822b876f. Epub 2011 Aug 4. PMID 21821517
- [Background] Vandepitte C, Gautier P, Xu D, Salviz EA, Hadzic A. Effective volume of ropivacaine 0.75% through a catheter required for interscalene brachial plexus blockade. Anesthesiology. 2013 Apr;118(4):863-7. doi: 10.1097/ALN.0b013e3182850dc7. PMID 23353796
- [Background] Cobcroft MD. Letter: Bilateral spread of analgesia with interscalene brachial plexus block. Anaesth Intensive Care. 1976 Feb;4(1):73. No abstract available. PMID 1252000
- [Background] Dooley J, Fingerman M, Melton S, Klein SM. Contralateral local anesthetic spread from an outpatient interscalene catheter. Can J Anaesth. 2010 Oct;57(10):936-9. doi: 10.1007/s12630-010-9360-y. Epub 2010 Jul 23. PMID 20652841
- [Background] Fredrickson MJ, Kilfoyle DH. Neurological complication analysis of 1000 ultrasound guided peripheral nerve blocks for elective orthopaedic surgery: a prospective study. Anaesthesia. 2009 Aug;64(8):836-44. doi: 10.1111/j.1365-2044.2009.05938.x. PMID 19604186
- [Background] Gologorsky E, Leanza RF. Contralateral anesthesia following interscalene block. Anesth Analg. 1992 Aug;75(2):311-2. doi: 10.1213/00000539-199208000-00046. No abstract available. PMID 1632560
- [Background] Gomez RS, Mendes TC. Epidural anaesthesia as a complication of attempted brachial plexus blockade using the posterior approach. Anaesthesia. 2006 Jun;61(6):591-2. doi: 10.1111/j.1365-2044.2006.04647.x. PMID 16704597
- [Background] Kumar A, Battit GE, Froese AB, Long MC. Bilateral cervical and thoracic epidural blockade complicating interscalene brachial plexus block: report of two cases. Anesthesiology. 1971 Dec;35(6):650-2. doi: 10.1097/00000542-197112000-00022. No abstract available. PMID 5124750
- [Background] Lombard TP, Couper JL. Bilateral spread of analgesia following interscalene brachial plexus block. Anesthesiology. 1983 May;58(5):472-3. doi: 10.1097/00000542-198305000-00016. No abstract available. PMID 6838002
- [Background] Fritsch G, Hudelmaier M, Danninger T, Brummett C, Bock M, McCoy M. Bilateral loss of neural function after interscalene plexus blockade may be caused by epidural spread of local anesthetics: a cadaveric study. Reg Anesth Pain Med. 2013 Jan-Feb;38(1):64-8. doi: 10.1097/AAP.0b013e318277a870. PMID 23222362
- [Background] Orebaugh SL, McFadden K, Skorupan H, Bigeleisen PE. Subepineurial injection in ultrasound-guided interscalene needle tip placement. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):450-4. doi: 10.1097/AAP.0b013e3181e859f0. PMID 20814286
- [Derived] Stundner O, Meissnitzer M, Brummett CM, Moser S, Forstner R, Kokofer A, Danninger T, Gerner P, Kirchmair L, Fritsch G. Comparison of tissue distribution, phrenic nerve involvement, and epidural spread in standard- vs low-volume ultrasound-guided interscalene plexus block using contrast magnetic resonance imaging: a randomized, controlled trial. Br J Anaesth. 2016 Mar;116(3):405-12. doi: 10.1093/bja/aev550. PMID 26865133